CLINICAL TRIAL: NCT00572104
Title: Efficacy of Plyometrics to Increase Bone Mass in Men With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1095877; R03AR055738 (NIH)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Resistance Training; Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resistance exercise (Experimental): 12 month resistance exercise training
  Interventions: Other: resistance exercise
- plyometric exercise (Experimental): 12 month plyometric exercise training
  Interventions: Other: plyometric exercise

INTERVENTIONS:
Other: resistance exercise — 12 month training intervention of weight resistance exercise. All participants receive a daily calcium and vitamin D supplement
  Arms: resistance exercise
Other: plyometric exercise — 12 month training intervention of plyometric exercise. All participants receive a daily calcium and vitamin D supplement
  Arms: plyometric exercise

SUMMARY:
This study will compare the ability of two types of long term (12 months) weight-bearing exercise treatments (1. high-intensity jumping and 2. weight lifting) to increase bone mass of the total body, spine and hip in physically active men with osteopenia.

DETAILED DESCRIPTION:
The overall goal of this project is to determine the efficacy of chronic (12 months) plyometric jump training exercise on bone mineral density (BMD) and markers of bone turnover in physically active males cyclists diagnosed with osteopenia below normal bone mineral density of the lumbar spine or hip.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 25-60 years
* No symptoms of disease
* Currently participating in cycling activities an average of 4 hr/wk for the previous 24 months
* Osteopenia of the lumbar spine and/or hip (T score < -1.0 and > -2.5 )

Exclusion Criteria:

* Medications or supplements that affect bone metabolism or prevent exercise
* Previous or current medical condition affecting bone health
* Osteoporosis of the lumbar spine and/or hip (T score > -1.0 or < -2.5)
* Cardiovascular disease
* Metallic implants
* Current smoker
* Current regular participation in high-intensity resistance training and/or plyometrics

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 12 months

SECONDARY OUTCOMES:
Serum markers of bone turnover | 3 months
Serum hormones regulating bone turnover | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela S Hinton, Principal Investigator — University of Missouri-Columbia, Department of Nutritional Sciences
Locations (1):
- University of Missouri-Columbia; McKee Gym, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No